CLINICAL TRIAL: NCT05139485
Title: Evaluation of a Remote Asthma Monitoring Program to Improve Health Outcomes in Pediatric Asthma
Status: Terminated | Type: Observational
Why Stopped: Staffing issues with partner site.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 20-06022311
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Asthma in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this pilot study to is to determine the overall impact of a clinical program of remote medication monitoring administered by St. Mary's Homecare on disease control in pediatric asthma patients. The central hypothesis is that a short-term program of remote asthma medication monitoring paired with home visits and asthma education will be associated with a sustained improvement in asthma symptom control in children over time.

DETAILED DESCRIPTION:
This is a pilot, prospective observational cohort study of 20 children with poorly controlled persistent asthma over 12 months exploring response to an intensive asthma monitoring and education program. The program consists of the following administered over a 6-month period: 1) A remote medication monitoring system (Propeller devices and monitoring administered by St. Mary's Healthcare) and 2) home visits by St. Mary's asthma nurses. The Propeller devices are electronic inhaler sensors which monitor the use of metered dose inhalers (as well as other medication delivery devices) and captures the date and time of use. This is an FDA approved device aimed at promoting asthma self-management in a cost-effective manner. The sensor stores and transmits information via Bluetooth to a paired wireless data transmitter, which sends the data to a secured server accessible by St. Mary's Healthcare.

The study will consist of two phases described below. Phase 1 (Months 1-6): Subjects are enrolled in the St. Mary's Healthcare home visiting and remote medication monitoring program through referral by the physicians/nurse practitioners providing asthma care and the Weill Cornell Pediatric Asthma Program. They will then undergo an initial home visit by a St. Mary's asthma program nurse, where they are equipped with Propeller devices for their controller medication (as prescribed by their physician) and rescue medication (albuterol), and are connected to St. Mary's remote monitoring system. Remote monitoring, home visits and in-person/video visit clinical assessment with asthma education will be provided during this time (see below). The St. Mary's remote monitoring system and telehealth nurse collects medication administration data obtained through the Propeller monitoring system in real-time, which is made available clinically to the subjects' medical providers on a monthly basis for review, or if there is substantial deviation from prescribed medication administration or increased use of rescue medication necessitating an intervention by St. Mary's telehealth nurses.

Additionally, the following outcomes data will be collected on a monthly basis via telephone or office/video visit by the study team to assess overall asthma control and health care use: Number of emergency room visits or hospitalizations for asthma in the last month, number of urgent care or primary care visits for asthma symptoms, number of albuterol prescriptions renewed, number of oral steroid prescriptions filled, number of missed school days, and an ACT score to assess control. Pulmonary function testing (PFT) will be performed at the time of enrollment.

Phase 2 (Months 7-12): Subjects will have completed remote asthma medication monitoring by the St. Mary's Program, and are observed for an additional 6 months by the study team to determine the response to the administered program. Subjects will have outcomes data (as described in Phase 1) collected via telephone or video visit; a minimum of 2 provider office or video visits will occur during this phase. PFTs will be performed at least once during this period.

Remote monitoring: Remote devices collect prospective data regarding use of controller medication as prescribed and any doses of rescue medication administered. If a patient is using their rescue inhaler above or using their controller inhaler less than prescribed, a St. Mary's Telehealth Nurse will receive an alert in real time. The Telehealth Nurse will contact the patient or caregiver to assess the situation and intervene, either by providing reminders or assessing for changes in clinical status. The Telehealth Nurse will initiate communication with their medical provider or emergency services as appropriate.

Home visits: Subjects enrolled in this program will be provided with up to 6 asthma nursing visits over the 12month study period as standard practice of St. Mary's home visitation program and based on the individual needs of the subject. A minimum of 2 nursing visits will be administered during phase 1 for clinical monitoring and asthma education/asthma management reinforcement.

Provider visits: Patients will have a physician office or video visit with NYPH-WCM providers scheduled during Month 2 and Month 5 of Phase 1 for standard clinical follow up, and to review their medication usage and provide directed feedback. This will be bundled with a dedicated asthma education session with WCM-Pediatric Asthma Program asthma educators to review/reinforce medication administration techniques and provide tailored asthma education for the development of asthma self-management skills. There will be a minimum of 2 scheduled Provider visits during Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 3- 21 years
* Diagnosis of persistent asthma (mild, moderate, severe) previously diagnosed by a physician
* Diagnosis of poorly controlled asthma or and asthma control test (ACT) score of <19

Exclusion Criteria:

* Patients who have severe cognitive delay, significant mental illness which impairs daily functioning or are non-verbal will be excluded as they are less likely to benefit from the educational techniques administered
* Primary language other than English or Spanish

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects between the ages of 3 and 21 years who have a diagnosis of persistent asthma (mild, moderate or severe) who have poorly controlled symptoms
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Change in asthma control test (ACT) scores | Baseline (enrollment), Month 6 and Month12
  This outcome will compare ACT scores at the time of enrollment, to month 6 and month 12 scores

SECONDARY OUTCOMES:
Change in percent of Controller Medication administered | 3 months, 6 months and 12months
  The percent of prescribed medication doses administered per month with comparison of mean percentage at month 3, month 6 and month 12
Change in number of Rescue Medication doses administered | 3 months, 6 months and 12months
  The number of rescue medication doses administered per month, with comparison of mean number of doses at month 3, month 6 and month 12
Change in health-care use: Number of physician visits | Enrollment, Month 12
  This secondary outcome will compare the number of physician visits due to asthma in the 12 month period pre-enrollment, to the number of physician visits due to asthma during the study period in month 12 (at completion of study).
Change in health-care use: Number of Emergency Department (ED) visits | Enrollment, Month 12
  This secondary outcome will compare the number of ED visits due to asthma in the 12 month period pre-enrollment, to the number of ED visits due to asthma during the study period in month 12 (at completion of study).
Change in health-care use: Number of Hospitalizations | Enrollment, Month 12
  This secondary outcome will compare the number of hospitalizations due to asthma in the 12 month period pre-enrollment, to the number of hospitalizations due to asthma during the study period in month 12 (at completion of study).
Change in health-care use: Number of oral steroid courses | Enrollment, Month 12
  This secondary outcome will compare the number of oral steroid courses prescribed due to an asthma exacerbation in the 12 month period pre-enrollment, to the number of oral steroid courses prescribed over the study period at month 12.
Change in number of missed school days | Enrollment, month 12
  Number of missed school days due to asthma in the 12-month period prior to enrollment compared to number of school days missed over the study period at month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Ono, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States